CLINICAL TRIAL: NCT07388576
Title: A Randomized, Triple-blind, Placebo-controlled, Parallel, Proof-of-concept Clinical Trial to Investigate the Safety and Efficacy of AP-Brain on Cognitive Function at Varying Dosages in Healthy Younger Adults With Self-reported Attention Problems
Brief Title: A Clinical Trial to Investigate the Safety and Efficacy of AP-Brain on Cognitive Function at Varying Dosages in Healthy Younger Adults With Self-reported Attention Problems
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rousselot BVBA (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25RBCCT03
Record Dates: First submitted 2026-01-27; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cognition; Cognitive Function
Keywords: memory; cognitive function; AP-Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AP-Brain (1g) (Experimental): AP-Brain (1g) contains 1 g of hydrolyzed collagen in a capsule
  Interventions: Dietary Supplement: AP-Brain (1g)
- AP-Brain (3g) (Experimental): AP-Brain (3 g) contains 3 g of hydrolyzed collagen in a capsule
  Interventions: Dietary Supplement: AP-Brain (3g)
- AP-Brain (5g) (Experimental): AP-Brain (5 g) contains 5 g of hydrolyzed collagen in a capsule
  Interventions: Dietary Supplement: AP-Brain (5g)
- Placebo (Placebo Comparator): Placebo consists of Silicified Microcrystalline Cellulose, magnesium stearate, Hydroxypropyl cellulose, and titanium dioxide
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AP-Brain (1g) — Participants will be instructed to take one dose (5 tablets) of the study product with a standardized meal during their in-clinic visit. This group will receive 1 APBrain capsule and 4 placebo capsules.
  Arms: AP-Brain (1g)
Dietary Supplement: AP-Brain (3g) — Participants will be instructed to take one dose (5 tablets) of the study product with a standardized meal during their in-clinic visit. This group will receive 3 APBrain capsules and 2 placebo capsules
  Arms: AP-Brain (3g)
Dietary Supplement: AP-Brain (5g) — Participants will be instructed to take one dose (5 tablets) of the study product with a standardized meal during their in-clinic visit. This group will receive 5 APBrain capsules and 0 placebo capsules
  Arms: AP-Brain (5g)
Dietary Supplement: Placebo — Participants will be instructed to take one dose (5 tablets) of the study product with a standardized meal during their in-clinic visit. This group will receive 0 AP-Brain capsules and 5 placebo capsules.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the safety and efficacy of AP-Brain on cognitive function at varying dosages in healthy younger adults with self-reported attention problems.

The main question it aims to answer is what Change from baseline to Day 56 between AP-Brain (1g, 3g, or 5g) and placebo in cognitive function, as assessed by the CNS VS Neurocognitive Index (NCI) score and complex attention.

Participants will be asked to consume AP-Brain at 1 g, 3 g, or 5g, or Placebo and asked to complete memory assessment questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18-39 years of age, inclusive
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active
3. Individuals with self-reported focus or attention problems, as determined by QI assessment of the Adult Attention Deficit Hyperactivity Disorder Self-Report Scale (Part A) (ASRS; version 1.1) (20)
4. Agrees to avoid high sources of caffeine (e.g., supplements, tea, coffee, energy drinks), NSAIDs, and alcohol consumption for 24 hours prior to post-screening clinic visits
5. Agrees to avoid first generation anti-allergy medication for 48 hours prior to post-screening clinic visits
6. Agrees to avoid moderate-vigorous exercise 12 hours prior to post-screening clinic visits
7. Agrees to avoid travel across two or more time zones two weeks prior to any study visit
8. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, and sleep) as much as possible throughout the study
9. Willing and able to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits
10. Provided voluntary, written, informed consent to participate in the study
11. Healthy as determined by medical history, laboratory results, and vital signs, as assessed by the QI

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product or placebo ingredients
3. Clinical diagnosis and/or prescribed treatment for ADHD (See Section 7.3.1)
4. Self-reported confirmation of any significant neuropsychological condition and/or cognitive impairment (e.g., Schizophrenia, bipolar disorder, post-traumatic stress disorder, brain injury, neurodegenerative disease, infections, insomnia, depression, epileptic or other seizure-related disorders) that could interfere with study participation as assessed by the QI
5. Self-reported color blindness/weakness as assessed by the QI
6. Individuals who consume high caffeine daily or are addicted to caffeine at screening as assessed by the QI
7. Current employment that calls for overnight shiftwork as assessed by the QI
8. Unstable metabolic disease or chronic diseases as assessed by the QI
9. Current or history of significant diseases of the gastrointestinal tract or conditions that result in malabsorption, as assessed by the QI
10. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI (See Section 7.3.1)
11. Type I diabetes
12. Type II diabetes if on insulin treatment. Type II diabetics on stable medication for at least three months and an HbA1c of <8.0% may be included after assessment by the QI on a case-by-case basis
13. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
14. History of or current diagnosis with kidney, gallbladder (e.g., gallstones, bile duct obstruction), and/or liver diseases (e.g., reduced bile salts, SIBO) as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
15. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
16. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
17. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
18. Individuals with an autoimmune disease or are immune compromised as assessed by the QI
19. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
20. Self-reported confirmation of blood/bleeding disorders as assessed by QI
21. Use of medical cannabinoid products
22. Chronic use of cannabinoid products (>2 times/week). Occasional users will be required to washout and abstain for the duration of the study period
23. Regular use of tobacco or nicotine products in the past six months, as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period
24. Alcohol intake average of >2 standard drinks per day as assessed by the QI
25. Alcohol or drug abuse within the last 12 months
26. Current use of prescribed and/or OTC medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the investigational product (Sections 7.3.1 and 7.3.2)
27. Clinically significant abnormal laboratory results at screening as assessed by the QI
28. Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the last study visit
29. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
30. Individuals who are cognitively impaired and/or unable to give informed consent
31. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Day 56 between AP-Brain and placebo in cognitive function, as assessed by the CNS VS Neurocognitive Index (NCI) score | Day 0 to 56
  Change from baseline to Day 56 between AP-Brain and placebo in cognitive function, as assessed by the CNS VS Neurocognitive Index (NCI) score and complex attention. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domain

SECONDARY OUTCOMES:
Change from baseline to Day 56 between AP-Brain and placebo in cognitive function, as assessed by complex attention via the CNS VS battery test | Day 0 to 56
  Change from baseline to Day 56 between AP-Brain and placebo in cognitive function, as assessed by complex attention. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in NCI Score as assessed by the CNS VS Neurocognitive Index (NCI) score. | Day 0 and 1
  Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: NCI Score. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in NCI Score assessed via CNS VS test battery. | Day 0 and 56
  Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: NCI Score. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in Complex attention via CNS VS test battery | Day 0 and 1
  Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Complex attention. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in Complex attention via CNS VS test battery | Day 0 and 56]
  Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Complex attention. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains
Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in Verbal, visual, composite, and working memory assessed via CNS VS test battery. | Day 0 and 1
  Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Verbal, visual, composite, and working memory. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in Verbal, visual, composite, and working memory assessed via CNS VS test battery. | Day 0 and 56]
  Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Verbal, visual, composite, and working memory. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains
Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Processing, motor, and psychomotor speed assessed via CNS VS test battery. | Day 0 and 1
  Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in Processing, motor, and psychomotor speed assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains
Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Processing, motor, and psychomotor speed assessed via CNS VS test battery. | Day 0 and 56
  Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Processing, motor, and psychomotor speed assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Reaction time assessed via CNS VS test battery. | Day 0 and 1]
  Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Reaction time assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Reaction time assessed via CNS VS test battery. | Day 0 and 56
  Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Reaction time assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Simple and sustained attention assessed via CNS VS test battery. | Day 0 and 1
  Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Simple and sustained attention assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Simple and sustained attention assessed via CNS VS test battery. | Day 0 and 56
  Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Simple and sustained attention assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domain
Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Executive function assessed via CNS VS test battery. | Day 0 and 1
  Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Executive function assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Executive function assessed via CNS VS test battery. | Day 0 and 56
  Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Executive function assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Cognitive flexibility assessed via CNS VS test battery. | Day 0 and 1
  Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Cognitive flexibility assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Cognitive flexibility assessed via CNS VS test battery. | Day 0 and 56
  Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Cognitive flexibility assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Impulsivity, defined as a composite score using reaction time, executive function, simple attention, and processing speed domains | Day 0 and 1
  Change from pre- to post-dose (t = 3h) at Days 1 between AP-Brain and placebo in the following CNS VS measures: Impulsivity, defined as a composite score using reaction time, executive function, simple attention, and processing speed domains assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Impulsivity, defined as a composite score using reaction time, executive function, simple attention, and processing speed domains. | Day 0 and 56
  Change from pre- to post-dose (t = 3h) at Days 56 between AP-Brain and placebo in the following CNS VS measures: Impulsivity, defined as a composite score using reaction time, executive function, simple attention, and processing speed domains assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change from baseline to Day 28 between AP-Brain and placebo in brain-derived neurotrophic factor (BDNF) Change from baseline to Day 28 between AP-Brain and placebo in brain-derived neurotrophic factor (BDNF) | Day 0 and 28
  Change from baseline to Day 28 between AP-Brain and placebo in brain-derived neurotrophic factor (BDNF) Change from baseline to Day 28 between AP-Brain and placebo in brain-derived neurotrophic factor (BDNF)
Change in cognitive function between AP-Brain and placebo based on the following measure: Change from baseline to Day 28 in CNS VS complex attention assessed via CNS VS test battery. | Day 0 and 28
  Change in cognitive function between AP-Brain and placebo based on the following measure: Change from baseline to Day 28 in CNS VS complex attention assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Verbal, visual, composite, and working memory assessed via CNS VS test battery. | Day 0 to 28
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Verbal, visual, composite, and working memory assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Verbal, visual, composite, and working memory assessed via CNS VS test battery. | Day 0 to 56
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Verbal, visual, composite, and working memory assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Processing, motor, and psychomotor speed assessed via CNS VS test battery. | Day 0 to 28
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Processing, motor, and psychomotor speed assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Processing, motor, and psychomotor speed assessed via CNS VS test battery. | Day 0 and 56
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Processing, motor, and psychomotor speed assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Reaction time assessed via CNS VS test battery. | Day 0 and 28
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Reaction time assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Reaction time assessed via CNS VS test battery. | Day 0 and 28
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Reaction time assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Simple and sustained attention assessed via CNS VS test battery. | Day 0 and 28
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Simple and sustained attention assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Simple and sustained attention assessed via CNS VS test battery. | Day 0 and 56
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Simple and sustained attention assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Executive function assessed via CNS VS test battery. | Day 0 and 28
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Executive function assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Executive function assessed via CNS VS test battery. | Day 0 and 56
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Executive function assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Cognitive flexibility assessed via CNS VS test battery. | Day 0 and 28
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Cognitive flexibility assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Cognitive flexibility assessed via CNS VS test battery. | Day 0 and 56
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Cognitive flexibility assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Impulsivity assessed via CNS VS test battery. | Day 0 and 28
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 28 in the following CNS VS measure: Impulsivity assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Impulsivity assessed via CNS VS test battery. | Day 0 and 56
  Change in cognitive function between AP-Brain and placebo based on change from baseline to Day 56 in the following CNS VS measure: Impulsivity assessed via CNS VS test battery. The CNS VS test battery is a validated cognitive assessment tool comprised of seven neurocognitive tests including a verbal and visual memory test, a finger tap test, symbol digit coding, the Stroop Test, a shifting attention test, and the continuous performance test. The CNS VS generates scores for the Neurocognitive Index which includes Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility, and for all individual domains.
Change between AP-Brain and placebo in insulin-like growth factor 1 (IGF-1) | Day 0 and 28
  Change between AP-Brain and placebo in insulin-like growth factor 1 (IGF-1)
Change between AP-Brain and placebo in insulin-like growth factor 1 (IGF-1) | Day 0 to 56
  Change between AP-Brain and placebo in insulin-like growth factor 1 (IGF-1)
Change between AP-Brain and placebo between AP-Brain and placebo in markers of inflammation, as assessed by Creactive protein (CRP), tumor necrosis factor alpha (TNF-α), and interleukin (IL)-6 | Day 0 to 28
  Change between AP-Brain and placebo between AP-Brain and placebo in markers of inflammation, as assessed by Creactive protein (CRP), tumor necrosis factor alpha (TNF-α), and interleukin (IL)-6
Change between AP-Brain and placebo between AP-Brain and placebo in markers of inflammation, as assessed by C-reactive protein (CRP), tumor necrosis factor alpha (TNF-α), and interleukin (IL)-6 | Day 0 to 56]
  Change between AP-Brain and placebo between AP-Brain and placebo in markers of inflammation, as assessed by C-reactive protein (CRP), tumor necrosis factor alpha (TNF-α), and interleukin (IL)-6
Difference in product perception between AP-Brain and placebo at Day 56, as assessed by the Product Perception Questionnaire (PPQ). | Day 0 to 56
  Difference in product perception between AP-Brain and placebo at Day 56, as assessed by the Product Perception Questionnaire (PPQ). Not scored on a scale, answers range from Strongly Agree to Strongly Disagree.

OTHER OUTCOMES:
Incidence of pre-emergent and post-emergent adverse events (AE) | Day 0 to 56
  Incidence of pre-emergent and post-emergent adverse events (AE)
Clinically relevant changes in vital signs (blood pressure (BP) after supplementation | Day 0 to 56
  Clinically relevant changes in vital signs (blood pressure (BP) after supplementation
Clinically relevant changes in heart rate (HR)) after supplementation | Day 0 to 56
  Clinically relevant changes in heart rate (HR)) after supplementation

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada